CLINICAL TRIAL: NCT00406900
Title: Melanoma Inhibitory Activity (MIA): A Serological Marker for Metastatic Uveal Melanoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Other Study IDs: MIA
Record Dates: First submitted 2006-11-29; First posted 2006-12-04 (Estimated); Last update posted 2006-12-06 (Estimated); Status verified 2006-11

CONDITIONS: Melanoma; Radiotherapy; Metastatic Disease
Keywords: uveal melanoma; metastatic disease
MeSH Terms: conditions — Melanoma; Neoplasm Metastasis; Uveal Melanoma

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Procedure: Treatment of metastatic disease

SUMMARY:
Uveal Melanoma is the most common primary intraocular tumor in adults. Most tumors metastasize to the liver. So far no sensitive or specific serological tumor marker is routinely used. The marker "Melanoma inhibitory activity" is a promising marker. Study hypothesis is to detect metastatic lesions in an early stage. This would increase life expectance of our patients

DETAILED DESCRIPTION:
Serum is taken from each melanoma patient at every follow up after signed concent. With ELISA the marker MIA is evaluated. An increase of MIA serum level will lead to search for metastasis by oncologists.

ELIGIBILITY:
Inclusion Criteria:

* uveal melanoma (With/without overt metastatic disease)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 560
Dates: Start 1999-01; Study Completion 2006-09

CONTACTS AND LOCATIONS:
Overall Officials: Ulrich C Schaller, MD, Principal Investigator — University of Munich, Germany
Locations (1):
- Dept of Ophthalmology, University of Munich, Munich, Germany

REFERENCES:
- [Result] Schaller UC, Bosserhoff AK, Neubauer AS, Buettner R, Kampik A, Mueller AJ. Melanoma inhibitory activity: a novel serum marker for uveal melanoma. Melanoma Res. 2002 Dec;12(6):593-9. doi: 10.1097/01.cmr.0000043146.28051.b8. PMID 12459649